CLINICAL TRIAL: NCT02888158
Title: Laparoscopic Training With and Without Robotic Assistance for Surgical Internes: a Randomized Study
Acronym: LAPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOI/2011/VL-01
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-08

CONDITIONS: Surgical Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic Trainer without robotic assistance (Active Comparator): Interns randomized to this arm will have two Pelvic Trainer training sessions three months apart.
  Intervention: Pelvic Trainer
  Interventions: Other: Pelvic Trainer
- Pelvic Trainer with robotic assistance (Experimental): Interns randomized to this arm will have two Pelvic Trainer training sessions three months apart but with robotic assistance.
  Intervention: Robotic assistance
  Intervention: Pelvic Trainer
  Interventions: Other: Robotic assistance; Other: Pelvic Trainer

INTERVENTIONS:
Other: Robotic assistance — Robotic assistance will be implemented during Pelvic Trainer training sessions.
  Arms: Pelvic Trainer with robotic assistance
Other: Pelvic Trainer — The standard Pelvic Trainer simulator for surgical training.

SUMMARY:
The primary objective of this study is to compare two groups of gynecologic/urologic/visceral internes in terms of the time required to perform a laparoscopic surgical intervention (nephrectomy) on an animal model (pig).

The two groups of internes differ by the type of training they received: (1) Pelvic-Trainer training with robotic assistance versus (2) Pelvic-Trainer training without robotic assistance.

ELIGIBILITY:
Inclusion Criteria:

* Intern registered for specialization in surgery (urological, visceral or gynecology-obstetrics)

Exclusion Criteria:

* The intern refuses to participate in the study
* The internal is not available for training and/or evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The time (in minutes) required for the intern to perform a laparoscopic nephrectomy on an animal model (pig). | 6 months (3 months after a second training session on the Pelvic Trainer)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Letouzey V, Huberlant S, Faillie JL, Prudhomme M, Mares P, de Tayrac R. Evaluation of a laparoscopic training program with or without robotic assistance. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:321-7. doi: 10.1016/j.ejogrb.2014.08.003. Epub 2014 Aug 20. PMID 25216348